CLINICAL TRIAL: NCT06703567
Title: IMproving PAtient UndeRstanding of GEP TEst Results: Phase 4
Acronym: IMPARTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IEO 1924
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Gene Expression Profiling; Oncotype DX
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): GEP test information (as per standard hospital policy)
  Interventions: Behavioral: Standard Policy
- GEP film (Experimental): Standard policy + the relevant GEP information film
  Interventions: Behavioral: Standard Policy + GEP Information Film

INTERVENTIONS:
Behavioral: Standard Policy — Patients will receive information about the GEP test by clinical teams
  Arms: Standard
Behavioral: Standard Policy + GEP Information Film — Patients will receive information about the GEP test by clinical teams and, after consultation with physician, they will be sent a link to view the film regarding OncotypeDX
  Arms: GEP film

SUMMARY:
The primary aim of the study is to determine if provision of a patient information film about Oncotype DX improves patients' knowledge and understanding about Gene Expression Profiling (GEP) test and risk of recurrence results in early breast cancer (EBC) patients, identified by their clinical teams as potentially benefiting from having their tumor samples sent for GEP analysis.

DETAILED DESCRIPTION:
Advances made in our understanding of the molecular biology of breast cancer have improved diagnostic testing and therapeutic options available to patients. Importantly results from genomic testing provide more accurate tailoring of treatments potentially enhancing the benefit to harm ratio by only offering adjuvant chemotherapy to those patients at highest risk of recurrence, and sparing those at lower risk the unwanted side effects of cytotoxic treatment. Conversations about risks and optimal treatments can be complex.

To aid understanding about GEP tests many clinical teams provide patients with information leaflets about GEP testing. Unfortunately these are often written by either academic or commercial sponsors and designed to meet certain ethical and regulatory guidelines rather than effectively educate the end-user.

There is some evidence that user-friendly patient information films might enhance patient knowledge and understanding and are more accessible to certain individuals, especially those with low literacy.

IMPARTER project has developed eight-minute film explaining why Oncotype DX GEP tests is used in EBC, what it is, and how the results help determine whether or not chemotherapy is recommended as a useful treatment option.

This study wish to examine the utility of the information film in the clinic setting with EBC patients identified by their clinical teams as potentially benefiting from having their tumor samples sent for GEP analysis.

ELIGIBILITY:
Inclusion Criteria:

* First presentation of early stage breast cancer with all known disease surgically removed
* Estrogen Receptor (ER) positive and Human Epidermal growth factor Receptor 2 (HER-2) negative
* No clear decision on whether chemotherapy should be given as adjunct based on current prognostic criteria
* Consented to GEP testing
* Able to give full informed consent to IMPARTER study
* Good comprehension of the Italian language
* Access to internet connection and devices (e.g. smart phone, tablet, laptop or desktop computer)

Exclusion Criteria:

* Other breast cancer diagnosis (e.g. Ductal carcinoma in situ, Metastatic)
* Unable to give fully informed consent
* Under 18 years of age
* Unable to understand and speak Italian
* No access to internet connection or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GEP Knowledge Evaluation | 1 week
  Collection of Gene Expression Profiling (GEP) Knowledge Questionnaire (higher total score indicates better understanding)

SECONDARY OUTCOMES:
Anxiety assessment | 1 week
  Collection of Spielberger State/Trait Anxiety Inventory (STAI) questionnaire (minimum value: 1, maximum value: 4 - higher scores signify greater anxiety)
Decision making assessment | 1 week
  Collection of Decisional Conflict Scale questionnaire (minimum value: 1, maximum value: 5 - higher scores mean a greater agreement with the statement)
Reaction to uncertain situations assessment | 1 week
  Collection of Intolerance of Uncertainty Scale Short-Form (IUS-12) questionnaire (minimum value: 1, maximum value: 5 - higher scores mean a greater agreement with the statement)
Physician confidence/satisfaction assessment | 1 week
  Collection of Confidence/satisfaction with GEP test result discussions questionnaire (higher scores indicate better satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy